CLINICAL TRIAL: NCT00901004
Title: Non-interventional, Cross-sectional, Multi-center Study to Establish The Clinical Significance of Minimal Change in Reflux Esophagitis Based on the Gastroesophageal Reflux Disease Questionnaire (GerdQ)
Brief Title: The Clinical Significance of Minimal Change in Reflux Esophagitis Based on the Gastroesophageal Reflux Disease Questionnaire
Acronym: MIGHT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-GKR-DUM-2009/1
Record Dates: First submitted 2009-04-28; First posted 2009-05-13 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Minimal Change; GERD; GERDQ
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Reflux esophageal minimal change in the endoscopic finding

SUMMARY:
The purpose of this study is to define the endoscopic findings of minimal change that is significant to clinical significant reflux esophagitis. Through this, the investigators want to estimate the applicability of minimal change findings of reflux esophagitis to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old patients who consent to revealing their medical information and be able to respond to questionnaires regarding the symptom.
* Patients who had shown the reflux esophageal minimal change in the endoscopic finding: the reflux esophagitis

Exclusion Criteria:

* Patients who had shown the mucosal break or barrett esophagus at gastric mucosal barrier or lower oesophagus in endoscopic findings
* Patient with a diagnosis of gastroesophageal reflux disease and who have received medication treatment
* Patient who had received H2-receptor antagonists, prostaglandin, PPI, NSAIDs or aspirin, high dose steroid and anticoagulants for at least 5 consecutive days in the 4-week period immediately preceding the diagnostic endoscopy
* Patients with a history of operation due to gastrointestinal disease, malignancy, alcoholism, pregnancy (in female), breast feeding (in female) or systemic disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had shown the reflux esophageal minimal change in the endoscopic finding
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Actual)
Dates: Start 2009-04; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To investigate significant minimal change endoscopic finding of reflux esophagitis diagnosis | Significant minimal change endoscopic finding for gastroesophageal reflux disease diagnosis

SECONDARY OUTCOMES:
To establish the probability model of diagnosing gastroesophageal reflux disease based on minimal change endoscopic findings through definition of significant minimal change endoscopic findings of gastroesophageal reflux disease diagnosis. | at baseline -->this is a cross-sectional study

CONTACTS AND LOCATIONS:
Overall Officials: Joonwoo Bahn, Study Director — Astrazenca Korea, Medical Department
Locations (7):
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejun
  - Research Site, Kwangju
  - Research Site, Seoul
  - Research Site, Sungman
  - Research Site, Suwon